CLINICAL TRIAL: NCT04180644
Title: Evaluation of Novel Skin Tape Transcriptome Methods in Children With Atopic Dermatitis and Healthy Controls
Brief Title: Skin Tape Transcriptome Methods in Children
Status: Completed | Type: Observational
Sponsor: National Jewish Health (Other)
Responsible Party: Sponsor
Other Study IDs: HS-3484
Record Dates: First submitted 2019-11-22; First posted 2019-11-27 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Atopic Dermatitis: Participants with atopic dermatitis active lesions
  Interventions: Other: Skin tape strips
- Healthy Control: Participants without a history of atopic dermatitis
  Interventions: Other: Skin tape strips

INTERVENTIONS:
Other: Skin tape strips — Skin tape strips will be collected from lesional and non-lesional skin. Adhesive skin sampling discs will be firmly pressed against the skin in a hairless location (not the face) followed by lifting it free of the skin. These discs will then be used to evaluate proteins and lipids in the upper layers of skin.

SUMMARY:
This pilot study will evaluate new methods for the collection, storage, shipment, and RNA extraction of skin tape specimens from children with atopic dermatitis (AD) that will facilitate the multi-center SunBeam Birth Cohort study. Additionally, this pilot study will test new methods for the generation of whole transcriptome sequencing data from skin tape RNA and whether these data reflect the transcriptional state of the skin in health and disease.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent/assent.
2. Male or female, 4-12 years of age (prepuberty) inclusive at the time of consenting
3. Participant must be either:

   1. Active atopic dermatitis with two areas of non-lesional AD within 5 cm of the measured lesional area within the same region.

      OR
   2. .No personal history or current manifestations of AD, food allergy, asthma, allergic rhinitis, and no positive prick or blood testing for allergen (based on self-report); and no evidence of dry skin or other skin condition

Exclusion Criteria:

1. Unable to provide consent or comply with the protocol
2. Presence of any skin condition that might compromise the stratum corneum barrier in infants and young children (e.g., ichthyosis, psoriasis, extensive seborrheic dermatitis, scabies)
3. History of any skin reaction to tape, or adhesives
4. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.
5. Use of any topical product (e.g., emollient, topical corticosteroids, topical immunomodulatory agents, topical antibiotics) on the area(s) to be tested within 24 hours before the study visit.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The investigators will recruit 20 children; 10 patients with moderate to severe AD and 10 healthy control subjects aged 4-12 (pre-puberty) years of age
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
skin RNA sequence for (lesional (L) and non-lesional (NL)) Skin Tape Strips (STS) | through study completion, single visit with an average of 2 hours
  the novel skin tape transcriptome method will extract RNA; the outcome is to identify the difference in RNA sequence between lesional and non-lesional skin.

CONTACTS AND LOCATIONS:
Locations (1):
- National Jewish Health and University of Colorado Denver, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No